CLINICAL TRIAL: NCT04500535
Title: A Multi-Center, Longitudinal, Prospective, Observational, Multi-Cohort Study of Patients With Advanced Non-Small Cell Lung Cancer Treated With Nivolumab in France After at Least One Prior Chemotherapy-based Treatment (LIST, Lung Initiative on Sequence Therapy)
Brief Title: A Study of Participants With Advanced Non-Small Cell Lung Cancer Treated With Nivolumab in France After at Least One Prior Chemotherapy-based Treatment by Lung Initiative on Sequence Therapy
Acronym: LIST
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-7HX
Record Dates: First submitted 2020-08-03; First posted 2020-08-05 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer
Keywords: Non Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Immuno-oncology (IO)-naïve patients
- Cohort 2: IO-experienced patients for whom last IO discontinuation was not primarily related to IO-toxicity
- Cohort 3: IO-experienced patients for whom last IO discontinuation was primarily due to IO-toxicity

SUMMARY:
The purpose of this trial is to describe the following, for each cohort, in real world conditions in France:

* The characteristics and treatment sequence of patients treated with nivolumab
* The effectiveness of nivolumab treatment
* The safety profile of nivolumab
* Treatment patterns (e.g. duration of treatment, subsequent treatments) of nivolumab
* The patient-reported outcomes (PRO) in patients treated with nivolumab, at baseline and during follow up using the EuroQoL-5D-3L

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Pathologically confirmed diagnosis of advanced NSCLC
* Whose physician has already decided to initiate a treatment with nivolumab for the treatment of advanced NSCLC according to the European label
* Previously treated with at least one prior chemotherapy- containing regimen

Exclusion Criteria:

* Participants taking part in an interventional study for lung cancer treatment for which nivolumab is one of the investigational drugs
* Participants with a diagnosis of another primary cancer within the past five years
* Participants receiving IO within 12 weeks prior to nivolumab first infusion in the context of the present study

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population will be constituted using multistage sampling, in which physicians (pulmonologists and/or oncologists) from eligible hospitals are to identify and recruit the participants. Eligible hospitals will be selected among PMSI sites (national hospital discharge database) and only hospitals with a minimum of 40 patients treated for lung cancer and with chemotherapy in 2018 will be considered to ensure sufficient enrollment.
Sampling Method: Probability Sample
Enrollment: 535 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure (TTF) | Up to 3 years

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 3 years
Progression-free survival (PFS) | Up to 3 years
Time to next therapy (TTNT) | Up to 3 years
Best overall response rate (BORR) | Up to 3 years
Distribution of participant demographics characteristics: Age | Index date (treatment initiation date for each individual patient
Distribution of participant demographics characteristics: Sex | Index date (treatment initiation date for each individual patient)
Distribution of clinical characteristics: Smoking status | Index date (treatment initiation date for each individual patient)
Distribution of clinical characteristics: ECOG at initial diagnosis and at nivolumab initiation | Index date (treatment initiation date for each individual patient)
Distribution of clinical characteristics: Histology | Index date (treatment initiation date for each individual patient)
Distribution of clinical characteristics: TNM classification | Index date (treatment initiation date for each individual patient)
  TNM=Tumor Nodes Metastases
Distribution of clinical characteristics: Location of metastases | Index date (treatment initiation date for each individual patient)
Distribution of clinical characteristics: EGFR mutation | Index date (treatment initiation date for each individual patient)
  EGRF=Epidural Growth Factor Receptor
Distribution of clinical characteristics: ALK translocation | Index date (treatment initiation date for each individual patient)
  ALK= Anaplastic Lymphoma Kinase
Distribution of clinical characteristics: HER2 mutation | Index date (treatment initiation date for each individual patient)
  HER2=Human Epidermal Growth Factor Receptor 2
Distribution of clinical characteristics: BRAF mutation | Index date (treatment initiation date for each individual patient)
Distribution of clinical characteristics: KRAS mutation | Index date (treatment initiation date for each individual patient)
Distribution of clinical characteristics: ROS1 mutation | Index date (treatment initiation date for each individual patient)
Distribution of clinical characteristics: MET mutation | Index date (treatment initiation date for each individual patient)
Distribution of clinical characteristics: PD-L1 expression | Index date (treatment initiation date for each individual patient)
  PD-L1=Programmed Death Ligand 1
Distribution of clinical characteristics: PD-L1 expression on tumor or stromal cells | Index date (treatment initiation date for each individual patient)
  PD-L1=Programmed Death Ligand 1
Incidence of Adverse Drug Reactions | 36 months after nivolumab treatment initiation
Incidence of Seriousness criteria | 36 months after nivolumab treatment initiation
Incidence of Intensity/ Grade | 36 months after nivolumab treatment initiation
Incidence of AE duration | Follow-up period (Week 4 to Week 156)
Incidence of Action taken regarding the BMS treatment | Follow-up period (Week 4 to Week 156)
Incidence of Incidence rate | Follow-up period (Week 4 to Week 156)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Paris, France

REFERENCES:
- [Derived] Godbert B, Gobbini E, Decroisette C, Lena H, Khalife Y, Brellier F, Fleuriet A, Zysman M, Egenod T, Moro Sibilot D, Girard N. Real-World Use and Immunotherapy Rechallenge Outcomes with Nivolumab in Advanced Non-small Cell Lung Cancer in France: Interim Results of the LIST Study. Oncol Ther. 2025 Dec;13(4):1071-1086. doi: 10.1007/s40487-025-00381-z. Epub 2025 Sep 14. PMID 40946253
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm